CLINICAL TRIAL: NCT00081380
Title: Multicenter, Randomized, Parallel-Group, Double-Blind, Phase 3 Comparison of the Efficacy & Safety of Quetiapine Fumarate to Placebo as Adjunct to Mood Stabilizers (Lithium or Divalproex) in the Maintenance Treatment of Bipolar I Disorder in Adult Patients (Abbreviated)
Brief Title: Efficacy and Safety of Seroquel Plus Mood Stabilizer in the Maintenance of Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D1447C00127
Record Dates: First submitted 2004-04-09; First posted 2004-04-19 (Estimated); Last update posted 2008-12-22 (Estimated); Status verified 2008-12

CONDITIONS: Bipolar Disorder
Keywords: Bipolar I Disorder; Manic Depressive Disorder; Manic Depression, Mixed
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate; Lithium; Valproic Acid

INTERVENTIONS:
Drug: Seroquel®, quetiapine fumarate (atypical antipsychotic)
Drug: lithium (mood stabilizer)
Drug: divalproex (mood stabilizer)

SUMMARY:
The purpose of this study is to determine whether quetiapine when used as adjunct to lithium or divalproex is safe and effective in the maintenance treatment of adult patients with Bipolar I Disorder. The study consists of enrollment and 2 phases, the Open-label treatment Phase and the Randomized treatment Phase.

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

Open-Label

* A diagnosis of Bipolar I Disorder, Most recent episode Manic (296.4x), or Bipolar I Disorder, Most Recent Episode Depressed (296.5x), or Bipolar I Disorder, Most recent Episode Mixed (296.6x), with or without psychotic features, as defined by Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition (DSM-IV)
* At least 1 manic, depressed, or mixed episode in the 2 years prior to the index episode.
* Able to understand and comply with the requirements of the study.

Exclusion Criteria:

Open-Label

* Diagnosis of an anxiety disorder as defined by DSM-IV, which was treated with medication within the past year.
* Known intolerance or lack of response to quetiapine fumarate or to the assigned mood stabilizer, as judged by the investigator.
* Previously randomized into this study or D1447C00126

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 710
Dates: Start 2004-03; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of quetiapine versus placebo when used as adjunct therapy to mood stabilizer in increasing time to recurrence of a mood event.

SECONDARY OUTCOMES:
Evaluate the efficacy of quetiapine versus placebo when used as a adjunct therapy to mod stabilizer in increasing time to recurrence of a manic event.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Seroquel Medical Science Director, MD, Study Director — AstraZeneca
Locations (94):
- United States (81):
  - Research Site, Birmingham, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Cerritos, California
  - Research Site, Chula Vista, California
  - Research Site, Culver City, California
  - Research Site, Garden Grove, California
  - Research Site, La Mesa, California
  - Research Site, Oceanside, California
  - Research Site, Orange, California
  - Research Site, Pico Rivera, California
  - Research Site, Riverside, California
  - Research Site, Rosemead, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Santa Ana, California
  - Research Site, Farmington, Connecticut
  - Research Site, New Britain, Connecticut
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Smyrna, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Chicago, Illinois
  - Research Site, Hoffman Estates, Illinois
  - Research Site, Joliet, Illinois
  - Research Site, Evansville, Indiana
  - Research Site, Greenwood, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Wichita, Kansas
  - Research Site, Florence, Kentucky
  - Research Site, Lake Charles, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Rockville, Maryland
  - Research Site, Pittsfield, Massachusetts
  - Research Site, New Baltimore, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Clementon, New Jersey
  - Research Site, Moorestown, New Jersey
  - Research Site, West Caldwell, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Brooklyn, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Butner, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Beachwood, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Medina, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Eugene, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Emmaus, Pennsylvania
  - Research Site, Moon Township, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, DeSoto, Texas
  - Research Site, Houston, Texas
  - Research Site, Irving, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Wichita Falls, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Falls Church, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Kirkland, Washington
  - Research Site, Morgantown, West Virginia
- Canada (13):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Halifax, Nova Scotia
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Markham, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec

REFERENCES:
- [Derived] Suppes T, Vieta E, Gustafsson U, Ekholm B. Maintenance treatment with quetiapine when combined with either lithium or divalproex in bipolar I disorder: analysis of two large randomized, placebo-controlled trials. Depress Anxiety. 2013 Nov;30(11):1089-98. doi: 10.1002/da.22136. Epub 2013 Jun 12. PMID 23761037